CLINICAL TRIAL: NCT05702749
Title: Evaluating Pre-Treatment Vestibular Physical Therapy Rehab for Patients with Vestibular Schwannomas
Acronym: VS PREHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael Harris, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00046306
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Vestibular Schwannoma
Keywords: stereotactic radiosurgery; Vestibular Schwannoma; sensory organization test
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Intervention: PREHAB and Surgery (Active Comparator): PREHAB exercises will be determined during the physical therapy visit (1x/week) and completed daily with varying frequency for three weeks. Subjects will undergo microsurgical resection of VS.
  Interventions: Procedure: Microsurgical resection of VS; Other: PREHAB
- Control: Surgery (No PREHAB) (Placebo Comparator): Subjects will undergo microsurgical resection of VS.
  Interventions: Procedure: Microsurgical resection of VS
- Intervention: PREHAB and SRS (Active Comparator): PREHAB exercises will be determined during the physical therapy visit (1x/week) and completed daily with varying frequency for three weeks. Subjects will undergo stereotactic radiosurgery.
  Interventions: Radiation: Stereotactic radiosurgery; Other: PREHAB
- Control: SRS (No PREHAB) (Placebo Comparator): Subjects will undergo stereotactic radiosurgery.
  Interventions: Radiation: Stereotactic radiosurgery

INTERVENTIONS:
Procedure: Microsurgical resection of VS — Microsurgical resection of VSs can be accomplished by three approaches including middle cranial fossa, retrosigmoid, and translabyrinthine. The surgical approach utilized is typically selected on the basis of tumor location and size, and patient age and hearing status.
  Arms: Control: Surgery (No PREHAB); Intervention: PREHAB and Surgery
Radiation: Stereotactic radiosurgery — Radiation therapy will be delivered using single fraction stereotactic radiosurgery with Gamma knife technology, or linear accelerator following institutional standard of care.
  Arms: Control: SRS (No PREHAB); Intervention: PREHAB and SRS
Other: PREHAB — A PREHAB visit will be done once weekly for 3 weeks to determine exercise regimen prior to surgery or radiotherapy. Therapy includes balance exercises (twice daily), gaze stabilization exercises (12-20 minutes daily), and habituation exercises (as applicable).
  Arms: Intervention: PREHAB and SRS; Intervention: PREHAB and Surgery

SUMMARY:
The study is a pilot efficacy study. The investigators aim to estimate mean baseline and post-treatment balance scores among Vestibular Schwannomas (VS) patients undergoing pretreatment rehab (PREHAB) or no PREHAB when managed with either surgery or radiosurgery.

DETAILED DESCRIPTION:
Study Design: This is a pilot randomized study with enrollment of 9 patients each to 4 groups: PREHAB+Surgery, No PREHAB+Surgery, PREHAB+Radiosurgery, and No PREHAB+Radiosurgery. Eighteen patients will be enrolled to receive each treatment type: surgery and radiosurgery. Within each type, patients will be randomized to PREHAB or NO PREHAB at a 1:1 ratio using stratified permuted blocks. The treatment modality will be determined by the patient and investigator(s) based upon collective consultations with neuro-otology, neurosurgery, and radiation oncology aligned with the Medical College of Wisconsin sporadic VS treatment guidelines.

Study Intervention: A PREHAB visit will be done once weekly for three weeks to determine exercise regimen prior to surgery or radiotherapy. Therapy includes balance exercises (twice daily), gaze stabilization exercises (12-20 minutes daily), and habituation exercises (as applicable). Standard surgical approaches including retrosigmoid, translabyrinthine, and middle fossa and radiosurgical (SRS) delivery will be determined based on current VS management guidelines and followed by study randomization to PREHAB.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male or female participants ≥18 years of age.
3. Initial diagnosis of a Vestibular Schwannoma confirmed by a physician with an internal auditory canal (IAC) MRI, in accordance with standard or institutional practice
4. VS patients who present with a tumor size ≤2.5 cm and will be treated with surgery or SRS
5. Eastern Cooperative Oncology Group (ECOG) Performance Status <2
6. Within 14 days of study registration, participants must have normal laboratory values that support safe treatment, at the discretion of the treating investigator
7. Be willing to adhere to outlined study protocol criteria and complete self-reported questionnaires (translations may be made available if the patient' primary language is not English).
8. For females of reproductive potential: must have a negative urine or serum pregnancy test 7 prior to enrollment and agreement to use of highly effective contraception method during study participation and for an additional 24 weeks after the completion of stereotactic radiosurgery.

Exclusion Criteria:

1. Subjects less than 18 years of age
2. Prior treatment of VS including radiotherapy or surgery or treatment for disease recurrence or planned salvage procedure
3. Pre-existing, secondary vestibular diagnoses (e.g., Meniere's, intractable benign paroxysmal positional vertigo (BPPV), vestibular migraine, 3PD).
4. Other medical comorbidities know to significantly impair/affect balance and/or vestibular function testing (e.g., prior stroke, uncorrected visual impairment or blindness, etc.)
5. Anticipated radiation other than stereotactic (fractionated)
6. Inability to undergo MRI scans safely
7. Allergy to Gadolinium contrast used for MRI scans
8. Women of childbearing potential who are known to be pregnant or are unwilling to use an acceptable method of contraception from the time of informed consent until completion of study related treatment and additional 24 weeks following stereotactic radiosurgery administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sensory Organization Test Score at Post-Treatment Assessments | Post-treatment 1 week
  The sensory organization test (SOT) was developed to describe the contribution levels of the three basic systems of balance (visual, vestibular, somatosensory) to the general equilibrium. The primary endpoint is the SOT at post-treatment assessments. This is measured by a composite score. A higher score equals greater stability. The measurement is made by a Bertec machine.
Sensory Organization Test Score at Post-Treatment Assessments | Post-treatment 6 weeks
  The sensory organization test (SOT) was developed to describe the contribution levels of the three basic systems of balance (visual, vestibular, somatosensory) to the general equilibrium. The primary endpoint is the SOT at post-treatment assessments. This is measured by a composite score. A higher score equals greater stability. The measurement is made by a Bertec machine.
Sensory Organization Test Score at Post-Treatment Assessments | Post-treatment six months
  The sensory organization test (SOT) was developed to describe the contribution levels of the three basic systems of balance (visual, vestibular, somatosensory) to the general equilibrium. The primary endpoint is the SOT at post-treatment assessments. This is measured by a composite score. A higher score equals greater stability. The measurement is made by a Bertec machine.
Sensory Organization Test Score at Post-Treatment Assessments | Post-treatment 12 months
  The sensory organization test (SOT) was developed to describe the contribution levels of the three basic systems of balance (visual, vestibular, somatosensory) to the general equilibrium. The primary endpoint is the SOT at post-treatment assessments. This is measured by a composite score. A higher score equals greater stability. The measurement is made by a Bertec machine.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitney SL, Marchetti GF, Schade AI. The relationship between falls history and computerized dynamic posturography in persons with balance and vestibular disorders. Arch Phys Med Rehabil. 2006 Mar;87(3):402-7. doi: 10.1016/j.apmr.2005.11.002. PMID 16500176
- [Background] Wrisley DM, Stephens MJ, Mosley S, Wojnowski A, Duffy J, Burkard R. Learning effects of repetitive administrations of the sensory organization test in healthy young adults. Arch Phys Med Rehabil. 2007 Aug;88(8):1049-54. doi: 10.1016/j.apmr.2007.05.003. PMID 17678669
- [Background] Hall CD, Herdman SJ, Whitney SL, Anson ER, Carender WJ, Hoppes CW, Cass SP, Christy JB, Cohen HS, Fife TD, Furman JM, Shepard NT, Clendaniel RA, Dishman JD, Goebel JA, Meldrum D, Ryan C, Wallace RL, Woodward NJ. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Updated Clinical Practice Guideline From the Academy of Neurologic Physical Therapy of the American Physical Therapy Association. J Neurol Phys Ther. 2022 Apr 1;46(2):118-177. doi: 10.1097/NPT.0000000000000382. PMID 34864777